CLINICAL TRIAL: NCT01915342
Title: Optimization of Physical Focal Stimulation Parameters for Improving Spasticity and Identification of Neurophysiological Mechanism
Brief Title: Developing Optimal Focal Muscle Vibration for Improving Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Institute of Science and Technology (Other)
Responsible Party: Principal Investigator, Byung-Mo Oh, Department of Rehabilitation Medicine, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FMV07-2013-1010
Record Dates: First submitted 2013-07-28; First posted 2013-08-02 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Vibration; Electrophysiology; Muscle Spasticity
Keywords: Monosynaptic reflex; H-reflex
MeSH Terms: conditions — Muscle Spasticity

ARMS (1):
- Focal muscle vibration (Experimental): Focal muscular vibration will be applied at mGCM of each subject for 10 minutes in each session.
  Frequency: 40, 80, 120 Hz Amplitude: 0.1, 0.3, 0.5 mm
  Interventions: Device: Focal muscular vibration

INTERVENTIONS:
Device: Focal muscular vibration

SUMMARY:
The overall aim of the proposed study is to determine optimal parameter of focal muscle vibration for improving spasticity and identify neurophysiological mechanism in healthy subjects.

In investigation I-1, subjects will undergo focal muscle vibration with 40, 80, 120 Hz frequency at the medial gastrocnemius muscles (mGCM). As a surrogate maker of spasticity, H-reflex and compound motor action potential (CMAP) of the tibial nerve at mGCM will be recorded pre, during, and post vibration.

In investigation I-2, subjects will undergo focal muscle vibration with 0.1, 0.3, 0.5 mm amplitude at mGCM. H-reflex and CMAP of the tibial nerve at mGCM will be recorded pre, during, and post vibration.

In investigation II, subjects will undergo focal muscle vibration with predetermined parameters by the investigation I at mGCM. H-reflex and CMAP of the tibial nerve and motor evoked potential at mGCM will be recorded pre, during, and post vibration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer

Exclusion Criteria:

* Unstable medical conditions
* History of epilepsy
* History of drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
H/M ratio | baseline, 1, 5 and 10 minutes during vibration, and 1 and 5 minutes after vibration
  The ratio of maximal H-reflex amplitude (mV) to CMAP amplitude (mV) recorded at mGCM

SECONDARY OUTCOMES:
H amplitude | baseline, 1, 5 and 10 minutes during vibration, and 1 and 5 minutes after vibration
  maximal H-reflex amplitude (mV) recorded at mGCM
M amplitude | baseline, 1, 5 and 10 minutes during vibration, and 1 and 5 minutes after vibration
  CMAP amplitude (mV) recorded at mGCM
motor evoked potential (MEP) amplitude | baseline, 10 minutes during vibration, and 5 minutes after vibration
  Transcranial magnetic stimulation on the contralateral leg motor cortex is used to measure MEP at mGCM.
Resting motor threshold (RMT) | baseline, 10 minutes during vibration, and 5 minutes after vibration
  Resting motor threshold (%) is defined as the minimal intensity of TMS capable of inducing MEPs greater than 100μV peak-to-peak amplitude in at least 3 of 5 trials.
Short interval intracortical inhibition | baseline, 10 minutes during vibration, and 5 minutes after vibration
  Short interval intracortical inhibition is recorded by using conditioning stimulus of 90% RMT and test stimulus of 120% RMT with 1ms interval.
Intracortical facilitation | baseline, 10 minutes during vibration, and 5 minutes after vibration
  Intracortical facilitation is recorded by using conditioning stimulus of 90% RMT and test stimulus of 120% RMT with 10ms interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea